CLINICAL TRIAL: NCT04908618
Title: Comparing the Accuracy of Intraoral Scanning of Ready Made Abutments Versus Intraoral Scan Bodies, Digitized Conventional Open and Closed Tray Implant Impression Techniques. A Controlled Clinical Trial
Brief Title: The Accuracy of Conventional Versus Digital Implant Impression Techniques
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mohamed Mahmoud Dohiem (Other Government)
Responsible Party: Sponsor-Investigator, Mohamed Mahmoud Dohiem, lecture prosthetic department zagazig university egypt, Zagazig University
Organization: Zagazig University (Other Government)
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 256413854
Record Dates: First submitted 2021-05-21; First posted 2021-06-01 (Actual); Last update posted 2021-06-01 (Actual); Status verified 2021-05

CONDITIONS: Missing Teeth
MeSH Terms: conditions — Anodontia

STUDY DESIGN:
Intervention Model Description: control clinical trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- digital impression with normal abutment for dental implant (Active Comparator): digital impression using a ready-made abutment for dental implant
  Interventions: Other: digital impression for normal abutment; Other: open tray impression; Other: closed tray impression
- digital impression with scan abutment for dental implant (Experimental): digital impression with scan body abutment for dental implant
  Interventions: Other: digital impression for normal abutment; Other: open tray impression; Other: closed tray impression
- open tray conventional dental implant impression (Experimental): Digitized open tray dental implant impression
  Interventions: Other: digital impression for normal abutment; Other: open tray impression; Other: closed tray impression
- closed tray impression for dental implant (Experimental): Digitized closed tray dental implant impression
  Interventions: Other: digital impression for normal abutment; Other: open tray impression

INTERVENTIONS:
Other: digital impression for normal abutment — Accuracy of scan body impression
Other: open tray impression — Accuracy of open tray impression
Other: closed tray impression — Accuracy of closed tray impression
  Arms: digital impression with normal abutment for dental implant; digital impression with scan abutment for dental implant; open tray conventional dental implant impression

SUMMARY:
Intraoral oral scanning significantly improves scanning accuracy compared to digitized conventional impression techniques. The digitized closed tray impression technique showed significantly more accurate results than the digitized open-tray impression technique in partially edentulous patients.

DETAILED DESCRIPTION:
The study was a controlled clinical trial using cone-beam computed tomography (CBCT) imaging and flapless surgical technique to place implants. Cone-beam Computed Topography of the patients was taken by x-ray machine to create a DICOM file of the patient. Intraoral scanning to create STL Files of the patient arches. Each patient had undergone four impression techniques: Conventional impression I; Closed tray impression technique, Conventional impression II; Splinted Open tray impression technique, Digital impression I; intraoral scanning of readymade abutments and Digital impression II; intraoral scanning using scan bodies. To digitize the Conventional impressions I and II, the readymade abutment was screwed on the analogs of the resultant stone casts, followed by digital scanning. Using the scan body, the exact implant position was determined and the implants were added using a digital library. The custom abutment was fabricated on the implant replica with the same readymade abutment measurement. Using the inspection software, a custom abutment was superimposed on each readymade abutment in all the readymade abutment scanning data with the best-fit algorithm. Then the custom abutment was saved as a new STL file for comparison. The digital impression I was set as a reference in all the coming comparisons. The comparison was done from different data acquisition techniques by using inspection software between Digital impression I, Digital impression II; and finally, with the digitized STL of the Conventional impressions I and II.

ELIGIBILITY:
Inclusion Criteria:

* Partial edentulous patients

  * Sufficient bone volume to insert implants
  * Age ranging from 30-50.
  * Good oral hygiene.
  * Intact hard and soft tissues, including treated teeth decay and healed teeth extraction socket

Exclusion Criteria:

* • Completely edentulous patients

  * Patients with Bruxism or clinching
  * need for bone augmentation,
  * uncompensated diabetes mellitus,
  * immunocompromised status, radio- and/or chemotherapy
  * previous treatment with oral and/or intravenous aminobisphosphonates.
  * Undergoing orthodontic treatment;
  * Patients with metal crowns and any other metal materials on teeth
  * Patients with soft tissue lesions and postoperative scars on the palate

Ages: 30 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Estimated)
Dates: Start 2021-05-20 (Actual); Primary Completion 2021-05-21 (Actual); Study Completion 2021-05-22 (Estimated)

PRIMARY OUTCOMES:
total deviation between digital impression and conventional impression | 1 day

CONTACTS AND LOCATIONS:
Locations (1):
- Mohamed Mahmoud Dohiem, Cairo, Egypt